CLINICAL TRIAL: NCT01901783
Title: Ridge Augmentation Comparing the Clinical and Histologic Healing of a Cancellous Block Allograft Plus a Barrier Membrane With and Without Primary Closure
Brief Title: Ridge Augmentation Without Primary Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.0331
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Alveolar Ridge Augmentation
Keywords: allograft; regeneration; alveolar ridge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- With primary closure (Active Comparator): The ridge augmentation graft will be covered with a barrier membrane and the soft tissue will be primarily closed.
  Interventions: Procedure: With primary closure
- Without primary closure (Experimental): The ridge augmentation graft will be covered with a barrier membrane and the soft tissue will not be primarily closed.
  Interventions: Procedure: Without primary closure

INTERVENTIONS:
Procedure: With primary closure — A cancellous block allograft will be placed for ridge augmentation and covered with a barrier membrane. The soft tissue will be primarily closed over the membrane.
  Other Names: Primary soft tissue closure over the membrane.
  Arms: With primary closure
Procedure: Without primary closure — A cancellous block allograft will be placed for ridge augmentation and covered with a barrier membrane. The soft tissue will not be primarily closed over the membrane.
  Other Names: No primary soft tissue closure over the membrane.
  Arms: Without primary closure

SUMMARY:
This study is designed to compare the clinical and histologic results of ridge augmentation with and without primary closure over the barrier membrane. The hypothesis is that there will be no difference in crestal ridge width between the two groups.

DETAILED DESCRIPTION:
A maximum of 30 patients will be selected that meet the following criteria:

Inclusion Criteria

1. At least a one tooth area with a ridge defect, treatment planned to receive a dental implant. The site must be bordered by at least one tooth.
2. Healthy person that is at least 18 years old.
3. Patient understands and signs an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria

1. Patients with debilitating systemic diseases, diseases that affect the periodontium, or psychological problems that would interfere with treatment.
2. Previous head and neck radiation or chemotherapy within the previous 12 months.
3. Patients with known allergy to any of the materials that will be used in the study.
4. Smokers.
5. Patients who need prophylactic antibiotics prior to dental procedures.
6. Patients on long-term steroid therapy or oral bisphosphonates > 3 years or any IV biosphosphonates.
7. Patients who are pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. At least a one tooth area with a ridge defect, treatment planned to receive a dental implant. The site must be bordered by at least one tooth.
2. Healthy person that is at least 18 years old.
3. Patient understands and signs an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, diseases that affect the periodontium, or psychological problems that would interfere with treatment.
2. Previous head and neck radiation or chemotherapy within the previous 12 months.
3. Patients with known allergy to any of the materials that will be used in the study.
4. Smokers.
5. Patients who need prophylactic antibiotics prior to dental procedures.
6. Patients on long-term steroid therapy or oral bisphosphonates > 3 years or any IV biosphosphonates.
7. Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Crestal ridge width | 4 months
  The ridge width at the crest will be compared between the two treatment groups.

SECONDARY OUTCOMES:
Percent vital bone | 4 months
  The percent vital bone will be compared between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic University of Louisville, Louisville, Kentucky, United States